CLINICAL TRIAL: NCT05960240
Title: A Double-Blind, Randomized, Placebo-Controlled, Single and Multiple Dose Study Evaluating the Safety, Tolerability, PK and PD of AB-101, an Oral PD-L1 Inhibitor, in Healthy Subjects and Subjects With Chronic HBV Infection.
Brief Title: Safety, Tolerability, PK & PD of AB-101 Following Oral Administration in Healthy and CHB Subjects.
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Arbutus Biopharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AB-101-001
Record Dates: First submitted 2023-07-14; First posted 2023-07-25 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1 (Experimental)
  Interventions: Drug: AB-101; Drug: Placebo
- Part 2 (Experimental)
  Interventions: Drug: AB-101; Drug: Placebo
- Part 3 (Experimental)
  Interventions: Drug: AB-101; Drug: Placebo; Drug: Nucleos(t)ide Analogue

INTERVENTIONS:
Drug: AB-101 — AB-101 is an oral small molecule PD-L1 checkpoint inhibitor being developed for the treatment of chronic infection with HBV in combination with other agents.
Drug: Placebo — A placebo is any treatment that has no active properties, such as a sugar pill. We will use matching placebo for this study.
Drug: Nucleos(t)ide Analogue — Nucleos(t)ide analogues (NUCs) are the standard and mostly lifelong treatment for chronic HBeAg-negative hepatitis B.
  Arms: Part 3

SUMMARY:
This three-part, Phase 1 protocol will be the first clinical study of AB-101. Parts 1 and 2 will be a Phase 1a SAD/MAD of AB-101 in healthy adult subjects.

Part 3 will be a Phase 1b dose-ranging assessment of AB-101 in non-cirrhotic Chronic Hepatitis B (CHB) subjects.

ELIGIBILITY:
Inclusion Criteria: Part 1 and 2 (Healthy Volunteers)

* Male between ages 18-50 years
* Willing and able to provide informed consent

Willing to follow protocol-specified contraception requirement

Inclusion Criteria: Part 3 (CHB Subjects)

* Male or female subjects between the ages of 18-60 years
* Willing to provide informed consent
* Chronic HBV infection for at least 6 months
* Willing to follow protocol-specified contraception requirement

Exclusion Criteria: Part 1 and 2 (Healthy Volunteers)

Key Exclusion Criteria:

* Clinically significant lab abnormalities
* A history of clinically significant gastrointestinal, hematologic, renal, hepatic, bronchopulmonary, neurological, psychiatric, cardiovascular, autoimmune or other immune-mediated disease.
* HIV or Hep C positive
* Known chronic or severe infection or recent significant exposure to infections such as tuberculosis or endemic mycosis, untreated latent infections like tuberculosis, or a positive or indeterminate QuantiFERON test.

Exclusion Criteria: Part 3 (CHB Subjects)

* Have extensive fibrosis or cirrhosis of the liver
* Have or had liver cancer (hepatocellular carcinoma)
* Have a history or current autoimmune disease or has been on immunosuppressive medications within 6 months of the start of the study
* Females who breastfeeding, pregnant or who wish to become pregnant during the study
* Known chronic or severe infection or recent significant exposure to infections such as tuberculosis or endemic mycosis, untreated latent infections like tuberculosis, or a positive or indeterminate QuantiFERON test.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Parts 1 and 2: Incidence of adverse events (AEs), serious AEs (SAEs), immune related AEs (irAEs) and discontinuations due to AEs and irAEs. | [Time Frame: Up to 57 (Part 1) or 84 (Part 2) days]
Part 3: Incidence of AEs, SAEs, irAEs and discontinuations due to AEs and irAEs | [Time Frame: Up to 196 days]
Parts 1 and 2: Incidence of clinically significant laboratory abnormalities Parts 1 and 2: Incidence of clinically significant laboratory abnormalities | [Time Frame: Up to 57 (Part 1) or 84 (Part 2) days]
Parts 1 and 2: Incidence of clinically significant changes in vital signs (heart rate, blood pressure, temperature, respiratory rate), physical examinations and electrocardiograms (ECGs) | [Time Frame: Up to 57 (Part 1) or 84 (Part 2) days]
Part 3: Incidence of clinically significant laboratory abnormalities | [Time Frame: Up to 196 days]
Part 3: Incidence of clinically significant changes in vital signs (heart rate, blood pressure, temperature, respiratory rate), physical examinations and electrocardiograms (ECGs) | [Time Frame: Up to 196 days]

CONTACTS AND LOCATIONS:
Locations (10):
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital - PPDS, Hong Kong
- Italy (2):
  - ASST Papa Giovanni XXIII -Osepedale, Bergamo
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
- Clinial Republican Hospital "Timofei Mosneaga", Chisinau, Moldova
- New Zealand Clinical Research Auckland, Grafton, Auckland, New Zealand
- Clinical Republican Hospital "Timofei Mosneaga", ARENSIA E. M., Bucharest, Romania
- Singapore (2):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
- Municipal Non-Profit Enterprise Kyiv City Clinical Hospital No12 Executive Body of Kyiv City Council, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided